CLINICAL TRIAL: NCT01449721
Title: Preemptive Empiric Resuscitation Protocol for the Prevention of Disease Progression in the Treatment of Sepsis
Brief Title: Preemptive Resuscitation for Eradication of Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRESHOCK
Record Dates: First submitted 2011-09-29; First posted 2011-10-10 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Sepsis; Severe Sepsis
Keywords: Sepsis; Multiple organ failure; Resuscitation
MeSH Terms: conditions — Sepsis; Multiple Organ Failure | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Standard medical care by the primary treatment team.
- Interventional arm (Experimental): Protocolized empiric resuscitation delivering weight-based intravenous fluid resuscitation targeting lactate normalization
  Interventions: Drug: Intravenous fluid

INTERVENTIONS:
Drug: Intravenous fluid — 0.9% Sodium chloride intravenous fluid
  Other Names: Normal saline
  Arms: Interventional arm

SUMMARY:
The purpose of this study is to assess the ability of an empiric resuscitation strategy compared to standard care to decrease the incidence of organ failure in normotensive sepsis patients.

DETAILED DESCRIPTION:
Sepsis is a challenging and elusive entity with a high mortality rate. As a syndrome, clinicians are challenged to distinguish individuals with systemic infection warranting further interventions from lower severity patients. Sepsis is now recognized as a time-sensitive emergency, as patients stand the best chance for survival when effective therapeutic interventions are delivered as early as possible.

Recent data has shown that in-hospital disease progression from sepsis to septic shock is associated with a higher risk of morbidity and mortality than those with shock on initial presentation. Yet, even when identified and treated with early aggressive interventions, the development of septic shock is still associated with a mortality rate of 25-40%.

Although the presence of sustained arterial hypotension or serum lactate elevation (>4.0 mmol/L) are the currently recommended threshold to define the presence of overt shock and the need for aggressive resuscitation, the investigators have shown that, in patients with systemic infection, a moderate lactate elevation (2.0-3.9 mmol/L) is a common occurrence and an important warning sign for the increased risk of disease progression and death. Sepsis with an elevated lactate between 2.0-3.9, referred to as the "PRE-SHOCK" state, identifies this population of patients at-risk for poor outcome. Current guidelines for sepsis management do not recommend any specific resuscitation measures or therapies for this at-risk population. This study marks the first in a series of investigations addressing the PRE-SHOCK population to further define the adverse events within this cohort and to investigate novel interventions to improve outcomes.

The investigators hypothesize that an early quantitative resuscitation strategy using a protocol-directed IV fluid resuscitation will result in a significant reduction in the development of worsening organ failure (including shock) and mortality compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Emergency department patient with suspected or confirmed infection as primary reason for admission
* Serum venous lactate 2.0 - 3.9 mmol/L
* Hospital admission planned

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Serum lactate ≥ 4.0 mmol/L
* Any vasopressor or inotrope requirement
* Mechanical ventilation or non-invasive positive pressure ventilation
* Chronic end-stage renal disease requiring hemodialysis
* Pulmonary edema as diagnosed by the primary care team
* Requirement for surgery within the treatment protocol timeframe
* Inability to obtain informed consent from subject or surrogate
* Patient to receive comfort measures only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2011-09; Primary Completion 2015-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Jones, MD, Study Chair — University of Mississippi Medical Center; Ryan Arnold, MD, Principal Investigator — Cooper University Hospital: Cooper Medical School of Rowan University
Locations (5):
- United States (5):
  - Christiana Care Health System, Newark, Delaware
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Detroit Receiving Hospital/University Health Center, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cooper University Hospital:Cooper Medical School of Rowan University, Camden, New Jersey

REFERENCES:
- [Background] Sakr Y, Vincent JL, Schuerholz T, Filipescu D, Romain A, Hjelmqvist H, Reinhart K. Early- versus late-onset shock in European intensive care units. Shock. 2007 Dec;28(6):636-643. PMID 18092378
- [Background] Mikkelsen ME, Miltiades AN, Gaieski DF, Goyal M, Fuchs BD, Shah CV, Bellamy SL, Christie JD. Serum lactate is associated with mortality in severe sepsis independent of organ failure and shock. Crit Care Med. 2009 May;37(5):1670-7. doi: 10.1097/CCM.0b013e31819fcf68. PMID 19325467
- [Background] Glickman SW, Cairns CB, Otero RM, Woods CW, Tsalik EL, Langley RJ, van Velkinburgh JC, Park LP, Glickman LT, Fowler VG Jr, Kingsmore SF, Rivers EP. Disease progression in hemodynamically stable patients presenting to the emergency department with sepsis. Acad Emerg Med. 2010 Apr;17(4):383-90. doi: 10.1111/j.1553-2712.2010.00664.x. PMID 20370777

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to interventional arm of the trial, a 5-month observational period was performed identifying 94 patients in the control arm. At the initiation of the interventional study, subjects were randomized in a 2:1 ratio to intervention:control, enrolling an additional 18 patients to the control arm, and 30 patients to the intervention.
Period: Overall Study
Arm/Group | Control | Interventional Arm
Started | 112 | 30
Completed | 112 | 28
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Interventional Arm | Total
Number analyzed (Participants) | 112 | 30 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (15) | 56.8 (16) | 58 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 12 | 63
  Male | 61 | 18 | 79

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Worsening Organ System Dysfunction Defined by SOFA Score Increase ≥ 1
Description: Development of worsening organ failure defined by the Sequential Organ Failure Assessment (SOFA) score. The SOFA score defines the presence and severity of dysfunction within 6 organ systems (cardiovascular, respiratory, coagulation, liver, renal, and nervous system) with a value of "0" for assigned to normal function to a maximum value of "4" for severe dysfunction in each of the organ systems. Each component of the SOFA score is added together, ranging from "0" indicating no organ dysfunction in any of the 6 organ systems, to "24" indicating maximal organ dysfunction across all 6 organ systems.
  Within this trial, the occurrence of organ failure was defined by any increase in the total SOFA score by ≥ 1 point over the first 72 hours after randomization.
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Interventional Arm
Number analyzed (Participants) | 112 | 30
Participants | 34 | 20
Statistical Analysis 1: Comparison: Control vs Interventional Arm; Null hypothesis: In patients with moderate severity sepsis, there is no change in the incidence of organ dysfunction within 72 hours associated with the use of an empiric fluid resuscitation algorithm; Test type: Superiority or Other; p = 0.064, 2-sample z-test; z-test for differences in proportions

2. Secondary Outcome: In-hospital Mortality
Description: Any occurrence of mortality while the participant is in-hospital is counted as an outcome.
Time Frame: In-hospital discharge or up to maximum 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Interventional Arm
Number analyzed (Participants) | 112 | 30
Participants | 4 | 0

3. Secondary Outcome: Number of Participants With Experiencing Complications Related to Intravascular Volume Overload
Description: Composite safety endpoint:
  * Premature termination of the protocol-directed intravenous fluid administration by the investigator or primary physician due to presumed volume overload
  * Administration of intravenous diuretic for acute pulmonary edema
  * Respiratory failure requiring ventilatory assistance (BiPAP, CPAP, or mechanical ventilation) secondary to pulmonary edema per primary care team
Time Frame: 12 hours following treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Interventional Arm
Number analyzed (Participants) | 112 | 30
Participants | 4 | 3

ADVERSE EVENTS:
Time Frame: Respiratory failure occurring within 24 hours of enrollment. Fluid overload occurring within 24 hours of enrollment. Mortality occurring at anytime within hospital stay.
Arm/Group | Control | Interventional Arm
All-Cause Mortality (participants affected / at risk) | 4/112 | 0/30
Serious Adverse Events (participants affected / at risk) | 4/112 | 3/30
Other Adverse Events (participants affected / at risk) | 0/112 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=112) | Interventional Arm (N=30)
Respiratory failure requiring mechanical intervention (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) — Any mechanical ventilation within 24 hours of enrollment.
Intravascular fluid overload (Vascular disorders) | 0 (0) | 2 (2) — Assessment by treating physician of intravascular fluid overload
Mortality (General disorders) | 4 (4) | 0 (0) — All cause in-hospital mortality

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No